CLINICAL TRIAL: NCT05881148
Title: Carbon " Super Spikes " Performances on Sprint Acceleration : Just Use it? A Multiple N-of-1 Trial. A Multiple N-of-1 Trial in Healthy Athletes
Brief Title: Carbon Sprinting Spiked-Shoes Trial
Acronym: CS3T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Léon Bérard (Other)
Responsible Party: Principal Investigator, Benjamin BERNUZ, MD, Dr Bernuz Benjamin; PMR; MD-MSc, Hôpital Léon Bérard
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2023-CS3T-Multiple N-of-1Trial
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Sprint Performance; Carbon Spiked-shoe; Force-velocity Profile; N of 1 Study Design

STUDY DESIGN:
Intervention Model Description: Multiple N-of-1 Trial: within-subjects repetitive blinded randomized crossovers
Who Masked: Participant, Outcomes Assessor
Masking Description: Each participant is self-blinded, but also blinded to other participants ' alternative order
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbon sprinting Super-spikes (Experimental): Trademarked Carbon Spiked-Shoes, from one Trademark only to ensure generalization concerns, is used alternatively with standard carbon-free spiked-shoes, for 8 repetitions of 30m-sprint each, separated by 10 minutes rest each.
  Interventions: Other: Carbon sprinting spiked-shoes
- Standard sprinting carbon-free spiked-shoe (Active Comparator)
  Interventions: Other: Standard carbon-free sprinting spiked-shoes

INTERVENTIONS:
Other: Carbon sprinting spiked-shoes — Trademarked Carbon Spiked-Shoes, from one Trademark only to ensure generalization concerns, is used alternatively with standard carbon-free spiked-shoes, for 8 repetitions of 30m-sprint each, separated by 10 minutes rest each.
  Other Names: carbon super-spikes
  Arms: Carbon sprinting Super-spikes
Other: Standard carbon-free sprinting spiked-shoes — cf
  Arms: Standard sprinting carbon-free spiked-shoe

SUMMARY:
Objectives :

To determine intra and inter-subject sprinting performance modifications with trademarked Carbon-made spiked-Shoes (CS) compared to usual carbon-free ones (Standard spiked-Shoes-SS).

Methods :

Design. Multiple N-of-1 trial (Alternating Treatments Design), with block randomisation and double blind procedure. For each participants, sixteen repetitions of 30m-sprint are applied either with CS or SS, in random order for each repetition, during a 3h session a day. Blind procedures are reached by applying a dark sleeve cover on each shoes, and by separating raters from investigators.

Patients. Regional to National healthy sprinting athletes (750 IAAF/WA points), affiliated to the French Athletics Federation among the South Regional Athletic League (Comité du Var-FFA), are recruited as volunteers, with their own CS (from the same brand for homogeneity and generalisation concerns) and SS.

Main criteria. Time on a 30-meters sprint, with Force-Velocity Profiling (FVP) procedure, using Stalker Sport radar.

Secondary outcome measures. F0, V0, Vmax, Pmax , DRP and other standard FVP parameters, also measured with MySprint software; morphometric and cinematic data ; mean price difference between the two models.

Statistical analyses. A block randomisation model will be applied to check for the randoms size; variance analysis with a mixt linear model will be applied for group and confounding factors analysis. Student-T test and NAP will be applied for intra-individuals analysis.

DETAILED DESCRIPTION:
Setting. The medical commission of the Var Athletics Committee (VAC), composed by medicine doctors, physiotherapists, universitary sport-scientists and FFA coaches, was in charge of the project, at Toulon conurbation and Draguignan, France.

Design. N-of-1 Trials is the usual term for randomized, double-blind SCEDs. This one has been designed as an Alternating Treatment Design (ATD), one of the four SCEDs types 25.

Due to the strict " on-off " intervention effect, no potential interference was expected between phases, and a " best treatment " final phase seems not necessary in the absence of carry-over or interaction effects. After discussion with coaches and athletes, the main constraint was to respect a single day " standard " short-sprint training session (i.e commonly 5 to 15 repetitions, up to 500m total volume). Respecting these conditions and the preference of athletes, ATD method seemed the more appropriate, allowing the most cycle comparisons in the same time span.

Procedure. For each participants, sixteen repetitions (2 sets of 8) of maximal 30m-sprint are applied, on the same track, either with " carbon super-spikes " (CS) or standard spikes (SS), in random order for each repetition, during a 3h total session a day. Repetitions are preceded by a full warm-up, and followed by a cool-down phase. Rest time between sets and repetitions is standardised (20 and 8-10 minutes).

Block starting can't be choosen in order to limit bias (reaction time, adjustment…) and to allow radar records at the pelvis height (1-m high), as recommended, so that a split-stance starting position was adopted, without any starter (" as soon as ready ").

A path is created between a " polling booth " zone, and the start- and finish lines. In this blinding zone, athletes are sitted on a wheelchair, blindfolded, and putted on with their shoes, which are already covered by dark socks allowing spikes free (athletes' visual blinding). Footwear management by the investigators avoid athletes to have tactile information (athletes'somesthesic blinding). Shoes can not be seen by raters (assessors' visual blinding) or other athletes in that zone. They are then driven to the start-line with the wheelchair, in order to limit gait sensation due to important differences in foams ± air-pods between CS and SS (athletes' proprioceptive blinding). This last point was added after athletes' contribution to the method.

At the start-line, they are asked for their belief between CS or SS, so that a " doubt " rate can be assessed to check for the blind paradigm. Then the blindfold is removed, and the subject stand-up in the starting position.

After the finish-line, a 20m deceleration zone is ended by a wheelchair, where athletes are blindfolded again, shoes tooken off and bringed back to the polling booth zone, as athletes enter the rest zone.

The wind is controlled with the official WA/FFA method and anemometer. The shoes weight is assessed, and standardised, when needed, with the addition of 20g ballasts glued at the heel, so that weight difference is decreased (<50g).

Data are collected and examined by two assessors blinded from the randomisation list.

Subjects. Healthy ≥ 15 years-old athletes presenting with a 750 IAAF/World Athletics points level in sprinting (60-400m), and affiliated to the VAC, are screened with the SIFFA software (Système d'Information-FFA). Fourty-six athletes are eligible, and are contacted by email, as their coaches, for information letter. Due to homogeneity and generalisation concerns, they have to have their own or lended Nike Zoom Maxfly or Victory style. Twenty-five respond positively, and N=21 are availables for one of the half-day-proposed sessions and are included.

ELIGIBILITY:
Inclusion Criteria:

* Sprinting athletes affiliated to the French Athletic Federation among the Var Athletics Comity
* Sprint Performance > 750pts IAAF/WA (50 to 400m)

Exclusion Criteria:

* Age<15
* Ongoing Injury

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-06-03 (Actual); Primary Completion 2023-08-06 (Actual); Study Completion 2023-08-06 (Actual)

PRIMARY OUTCOMES:
30m-sprint Time | in a 3 hour session a day
  16 x30m-sprint per subject

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Leon Berard, Hyères, Var, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request. For the Editorial office of the corresponding relevant editor; for meta-analyses needs, or for other detailed requests.
  From all types, with de-identified files (Morphometric, cinematic and FVP data, Statistical Analysis, etc..).
  Via a controlled access repositories, such as clinicalstudydatarequest.com, the YODA project, or Vivli.
Supporting Information: Study Protocol, SAP
Time Frame: as soon as leading article is published
Access Criteria: cf Plan Description

REFERENCES:
- [Background] Samozino P, Rabita G, Dorel S, Slawinski J, Peyrot N, Saez de Villarreal E, Morin JB. A simple method for measuring power, force, velocity properties, and mechanical effectiveness in sprint running. Scand J Med Sci Sports. 2016 Jun;26(6):648-58. doi: 10.1111/sms.12490. Epub 2015 May 21. PMID 25996964
- [Background] Edouard P, Lahti J, Nagahara R, Samozino P, Navarro L, Guex K, Rossi J, Brughelli M, Mendiguchia J, Morin JB. Low Horizontal Force Production Capacity during Sprinting as a Potential Risk Factor of Hamstring Injury in Football. Int J Environ Res Public Health. 2021 Jul 23;18(15):7827. doi: 10.3390/ijerph18157827. PMID 34360125
- [Background] Nagahara R, Kanehisa H, Fukunaga T. Influence of shoe sole bending stiffness on sprinting performance. J Sports Med Phys Fitness. 2018 Dec;58(12):1735-1740. doi: 10.23736/S0022-4707.17.07834-3. Epub 2017 Oct 27. PMID 29083127
- [Derived] Bernuz B, Laujac S, Sirial C, Auffret S, Preda C, Slawinski J, Millot B, Pradon D, Coudrat L, Gavarry O. Effect of Advanced Footwear Technology Spikes on Sprint Acceleration: A Multiple N-of-1 Trial. Sports Med Open. 2024 Aug 30;10(1):92. doi: 10.1186/s40798-024-00758-w. PMID 39214886